Version date: 12/10/2017 **Research Subject Informed Consent Signature Page** Title of Study: Implementing a Participatory, Multi-level Intervention to Improve Asian American Health Study # s17-01077 Mary E. Northridge, PhD, MPH (NYU College of Dentistry) **Principal Investigator:** have have not received and read the accompanying "Research Subject Informed Consent Brochure" Continue Below **ONLY** if you received and read the brochure. 14. Optional permission for future use NYULMC would also like to store, use, and share your health information from this study in research databases or registries for future research conducted by NYULMC or its research partners. Such health information may include biological samples from the study. To give this additional permission, check the box below and write your initials where indicated. You may still participate in this study even if you do not give us this additional permission. NYULMC will continue to protect the confidentiality and privacy of this information as required by law and our institutional polices. If you give this additional permission, you will continue to have the rights described in this form. You have the right to take back this additional permission at any time. Checking this box indicates my permission to store, use, and share my health information from this study in research databases or registries for future research conducted by NYULMC or its research partners. Subject Initials 15. The Institutional Review Board (IRB) and how it protects you The IRB reviews all human research studies - including this study. The IRB follows Federal Government rules and guidelines designed to protect the rights and welfare of the people taking part in the research studies. The IRB also reviews research to make sure the risks for all studies are as small as possible. The NYU IRB Office number is (212) 263-4110. The NYU School of Medicine's IRB is made up of: Doctors, nurses, non-scientists, and people from the Community 16. Who can I call with questions, or if I'm concerned about my rights as a research subject? If you have guestions, concerns or complaints regarding your participation in this research study or if you have any guestions about your rights as a research subject, you should speak with the Principal Investigators listed on top of the page 1 of this consent form. If a member of the research team cannot be reached or you want to talk to someone other than those working on the study, you may contact the NYU Institutional Review Board (IRB) at (212) 263-4110. When you sign this form, you are agreeing to take part in this research study as described to you. This means that you have read the consent form, your questions have been answered, and you have decided to volunteer. Name of Subject (Print) Signature of Subject Date Name of Person Obtaining Consent (Print) Signature of Person Obtaining Consent Date

## Statement of Witness I represent that the consent form was presented orally to the subject in the subject's own language, that the subject was given the opportunity to ask questions, and that the subject has indicated his/her consent and authorization for participation by (check box that applies): Subject making his/her own "X" above in the subject signature line Subject showed approval for participation in another way; describe:

Signature of Witness

Date

Witness to Consent of a Subject Who Cannot Read or Write

Name of Witness (Print)